CLINICAL TRIAL: NCT02915978
Title: A Phase 2 Multicenter, Randomized, Double-Blind, Multiple-Dose, Parallel-Group, Placebo-Controlled Study of Fentanyl Sublingual Spray for the Treatment of Moderate to Severe Post-Operative Pain
Brief Title: Fentanyl Sublingual Spray for the Treatment of Moderate to Severe Post-Operative Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS002-16-092
Record Dates: First submitted 2016-09-23; First posted 2016-09-27 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower Dose Fentanyl (Experimental): Lower dose Fentanyl delivered via sublingual spray every 4 hours.
  Interventions: Drug: Fentanyl
- Higher Dose Fentanyl Sublingual Spray (Experimental): Higher dose Fentanyl delivered via sublingual spray every 4 hours.
  Interventions: Drug: Fentanyl
- Placebo (Placebo Comparator): Placebo (matching Fentanyl) delivered via sublingual spray every 4 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl — Fentanyl delivered via sublingual spray
  Arms: Higher Dose Fentanyl Sublingual Spray; Lower Dose Fentanyl
Drug: Placebo — Matching placebo delivered via sublingual spray
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to evaluate analgesic efficacy of Fentanyl Sublingual Spray compared with placebo in participants with postoperative pain after a bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related to food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* History or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (2):
- United States (2):
  - Arizona Research Center, Phoenix, Arizona
  - Anaheim Clinical Trials, Anaheim, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (matching Fentany) delivered via sublingual spray every 4 hours.
  Placebo: Matching placebo delivered via sublingual spray
Period: Overall Study
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl | Placebo
Started | 15 | 15 | 15
Completed | 13 | 14 | 15
Not Completed | 2 | 1 | 0
Not completed — Adverse Event | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lower Dose Fentanyl Sublingual Spray: Lower dose Fentanyl delivered via sublingual spray every 4 hours.
  Fentanyl: Fentanyl delivered via sublingual spray
- Total: Total of all reporting groups
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (14.3) | 50.0 (10.6) | 45.5 (11.4) | 46.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 14 | 38
  Male | 3 | 3 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3 | 6
  Not Hispanic or Latino | 13 | 14 | 12 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 4 | 14
  White | 11 | 9 | 9 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Summed Pain Intensity Difference (SPID) Over 0 to 48 Hours (NRS SPID-48) After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points up to 48 hours after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum(max)=10 at each time point], and negative numbers indicate an increase in pain [minimum(min)=-10 at each time point]. The overall min and max are -10 and 10 times the number of hours specified; SPID-48 range is -480 to 480. The NRS SPID-48 was analyzed using an analysis of covariance (ANCOVA) model, which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Over 0 to 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
units on a scale | 151.7 (95.52) | 126.4 (124.66) | 149.0 (115.26)

2. Secondary Outcome: NRS Pain Intensity Difference (NRS PID) at Each Categorical Time Point After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug administration) and at multiple time points after Time 0 (time of administration of the first dose of study drug). NRS PID is defined as the difference in pain at each scheduled time point relative to Baseline (PID=pain intensity at baseline - pain intensity at time point). A higher value of NRS PID score indicates a higher decrease in pain from Baseline. NRS PID is reported as the least squares mean difference.
Time Frame: Baseline, 1, 16, and 24 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline | 6.5 (1.64) | 6.1 (2.13) | 7.1 (2.22)
  1 Hour | 3.7 (2.46) | 4.3 (2.09) | 5.8 (2.96)
  16 Hours | 2.6 (2.18) | 3.9 (3.04) | 5.5 (2.23)
  24 Hours | 2.0 (1.96) | 3.2 (2.21) | 3.3 (2.64)
Statistical Analysis 1: Comparison: Higher Dose Fentanyl Sublingual Spray vs Placebo; NRS PID at 1 hour; Test type: Other; p = 0.0505, ANCOVA; LS Mean Difference = -1.80, 95% CI 2-sided [-3.61 to 0.00], Standard Error of Mean 0.89
Statistical Analysis 2: Comparison: Lower Dose Fentanyl Sublingual Spray vs Placebo; NRS PID at 1 hour; Test type: Other; p = 0.2493, ANCOVA; LS Mean Difference = -1.06, 95% CI 2-sided [-2.89 to 0.77], Standard Error of Mean 0.90
Statistical Analysis 3: Comparison: Higher Dose Fentanyl Sublingual Spray vs Placebo; NRS PID at 16 hours; Test type: Other; p = 0.0052, ANCOVA; LS Mean Difference = -2.94, 95% CI 2-sided [-4.95 to -0.94], Standard Error of Mean 0.99
Statistical Analysis 4: Comparison: Lower Dose Fentanyl Sublingual Spray vs Placebo; NRS PID at 16 hours; Test type: Other; p = 0.0926, ANCOVA; LS Mean Difference = -1.67, 95% CI 2-sided [-3.62 to 0.29], Standard Error of Mean 0.97
Statistical Analysis 5: Comparison: Higher Dose Fentanyl Sublingual Spray vs Placebo; NRS PID at 24 hours; Test type: Other; p = 0.0951, ANCOVA; LS Means Difference = -1.40, 95% CI 2-sided [-3.06 to 0.26], Standard Error of Mean 0.82
Statistical Analysis 6: Comparison: Lower Dose Fentanyl Sublingual Spray vs Placebo; NRS PID at 24 hours; Test type: Other; p = 0.9866, ANCOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-1.60 to 1.63], Standard Error of Mean 0.80

3. Secondary Outcome: NRS Pain Intensity Score at Each Scheduled Time Point After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug administration) and at multiple time points after Time 0 (time of administration of the first dose of study drug). A lower value indicates improvement in pain.
Time Frame: Baseline, 1, 16, and 24 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Baseline | 6.5 (1.64) | 6.1 (2.13) | 7.1 (2.22)
  1 Hour | 3.7 (2.46) | 4.3 (2.09) | 5.8 (2.96)
  16 Hours | 2.6 (2.18) | 3.9 (3.04) | 5.5 (2.23)
  24 hours | 2.0 (1.96) | 3.2 (2.21) | 3.3 (2.64)

4. Secondary Outcome: NRS SPID After Time 0
Description: Pain intensity was assessed by the participant using an 11-point NRS from 0=no pain to 10=worst possible pain. Pain intensity scores were collected at Baseline (prior to study drug) and at multiple time points after Time 0 (administration of first dose of study drug). Pain intensity difference is calculated by subtracting the pain intensity at each time point from the pain intensity at Time 0. The SPID scores are the sum of the differences at each time point multiplied by the duration in hours since the previous time point. Positive numbers indicate a reduction in pain [maximum(max)=10 at each timepoint], and negative numbers indicate an increase in pain [minimum(min)=-10 at each timepoint]. The overall min and max are -10 and 10 times the number of hours specified: SPID-4=(-40 to 40), SPID-8=(-80 to 80) and SPID-24=(-240 to 240). The NRS SPID-4, 8 and 24 were analyzed using an ANCOVA model which included treatment and site as main effects and Baseline pain intensity as the covariate.
Time Frame: Over 0 to 4 hours (NRS SPID-4), over 0 to 8 hours (NRS SPID-8), and over 0 to 24 hours (NRS SPID-24)
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Over 24 Hours | 67.4 (40.45) | 51.7 (53.43) | 51.7 (59.38)
  Over 8 Hours | 13.6 (14.59) | 11.2 (16.18) | 8.8 (19.70)
  Over 4 Hours | 6.6 (7.58) | 5.9 (8.79) | 4.8 (12.73)

5. Secondary Outcome: Total Pain Relief (TOTPAR) After Time 0
Description: TOTPAR was assessed by the participant using a 5-point NRS (0=no relief, 1=a little, 2=some, 3=a lot, 4=complete relief). TOTPAR scores were collected at Baseline (prior to study drug) and at multiple time points up to 48 hours after Time 0 (first dose of study drug). The TOTPAR scores are the sum of the pain relief at each time point multiplied by the duration in hours since the previous time point. Larger positive numbers indicate more pain relief (maximum=4 at each time point) and smaller positive numbers indicate less pain relief (minimum=0 at each time point). The overall minimum is 0 for each variable and the overall maximum is 4 times the number of hours specified for the variable: TOTPAR-4=(0 to 16), TOTPAR-8=(0 to 32), TOTPAR-24=(0 to 96) and TOTPAR-48=(0 to 192). TOTPAR-4, TOTPAR-8, TOTPAR-24 and TOTPAR-48 were analyzed using an ANCOVA model with factors for treatment, site and baseline pain intensity.
Time Frame: Over 0 to 4 hours (TOTPAR-4), over 0 to 8 hours (TOTPAR-8), over 0 to 24 hours (TOTPAR-24), and over 0 to 48 hours (TOTPAR-48)
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
units on a scale
  Over 48 Hours | 98.2 (55.25) | 99.9 (33.63) | 98.2 (33.32)
  Over 24 Hours | 43.8 (22.72) | 46.5 (16.87) | 38.3 (14.81)
  Over 8 Hours | 11.6 (8.53) | 10.6 (6.32) | 7.2 (5.33)
  Over 4 Hours | 5.3 (4.54) | 5.1 (3.77) | 3.9 (4.53)

6. Secondary Outcome: Time to Onset of Analgesia
Description: Measured as time to perceptible pain relief confirmed by meaningful pain relief using the 2-stopwatch method (2 stopwatches will be started as soon as the first dose of study drug is administered. Each participant will be instructed to stop the first stopwatch when he or she experiences any perceptible pain relief and the second stopwatch when he or she experiences pain relief that is meaningful to them.)
Time Frame: Within 48 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
minutes | 5 [2 to 16] | 184 [1 to NA] — Not estimable because less than 50% of participants achieved onset. | NA [4 to NA] — Not estimable because less than 50% of participants achieved onset.

7. Secondary Outcome: Pain Relief at Each Scheduled Time Point After Time 0 (First Dose of Study Medication)
Description: Pain relief is determined on a 5-point categorical scale where 0=none, 1=a little, 2=some, 3=a lot, 4=complete.
Time Frame: 2.5, 5, 15, 30, and 45 minutes, and 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 16, 20, 24, 32, 40, and 48 hours, as well as immediately before each use of rescue analgesia
Population: All randomized participants from the Intent-to-Treat (ITT) population. The number analyzed differs in the later time points for the Fentanyl groups because some participants withdrew over the course of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
Participants
  2.5 Minutes After Time 0: No Relief | 9 | 9 | 11
  2.5 Minutes After Time 0: A Little Relief | 4 | 3 | 2
  2.5 Minutes After Time 0: Some Relief | 1 | 3 | 1
  2.5 Minutes After Time 0: A Lot of Relief | 1 | 0 | 1
  2.5 Minutes After Time 0: Complete Relief | 0 | 0 | 0
  5 Minutes After Time 0: No Relief | 6 | 9 | 10
  5 Minutes After Time 0: A Little Relief | 6 | 3 | 2
  5 Minutes After Time 0: Some Relief | 2 | 2 | 2
  5 Minutes After Time 0: A Lot of Relief | 1 | 1 | 1
  5 Minutes After Time 0: Complete Relief | 0 | 0 | 0
  15 Minutes After Time 0: No Relief | 5 | 3 | 9
  15 Minutes After Time 0: A Little Relief | 3 | 9 | 3
  15 Minutes After Time 0: Some Relief | 2 | 2 | 1
  15 Minutes After Time 0: A Lot of Relief | 5 | 1 | 1
  15 Minutes After Time 0: Complete Relief | 0 | 0 | 1
  30 Minutes After Time 0 - No Relief: No Relief | 3 | 3 | 9
  30 Minutes After Time 0 - No Relief: A Little Relief | 4 | 6 | 2
  30 Minutes After Time 0 - No Relief: Some Relief | 1 | 4 | 1
  30 Minutes After Time 0 - No Relief: A Lot of Relief | 5 | 2 | 2
  30 Minutes After Time 0 - No Relief: Complete Relief | 2 | 0 | 1
  45 Minutes After Time 0: No Relief | 3 | 4 | 7
  45 Minutes After Time 0: A Little Relief | 6 | 4 | 5
  45 Minutes After Time 0: Some Relief | 1 | 4 | 0
  45 Minutes After Time 0: A Lot of Relief | 2 | 3 | 1
  45 Minutes After Time 0: Complete Relief | 3 | 0 | 2
  1 Hour After Time 0: No Relief | 3 | 5 | 6
  1 Hour After Time 0: A Little Relief | 5 | 3 | 5
  1 Hour After Time 0: Some Relief | 3 | 4 | 2
  1 Hour After Time 0: A Lot of Relief | 2 | 3 | 0
  1 Hour After Time 0: Complete Relief | 2 | 0 | 2
  1.5 Hours After Time 0: No Relief | 5 | 4 | 6
  1.5 Hours After Time 0: A Little Relief | 4 | 3 | 2
  1.5 Hours After Time 0: Some Relief | 2 | 4 | 5
  1.5 Hours After Time 0: A Lot of Relief | 3 | 4 | 0
  1.5 Hours After Time 0: Complete Relief | 1 | 0 | 2
  2 Hours After Time 0: No Relief | 7 | 6 | 7
  2 Hours After Time 0: A Little Relief | 3 | 3 | 4
  2 Hours After Time 0: Some Relief | 0 | 3 | 2
  2 Hours After Time 0: A Lot of Relief | 4 | 3 | 0
  2 Hours After Time 0: Complete Relief | 1 | 0 | 2
  3 Hours After Time 0: No Relief | 7 | 5 | 7
  3 Hours After Time 0: A Little Relief | 3 | 4 | 3
  3 Hours After Time 0: Some Relief | 1 | 4 | 2
  3 Hours After Time 0: A Lot of Relief | 2 | 2 | 2
  3 Hours After Time 0: Complete Relief | 2 | 0 | 1
  4 Hours After Time 0: No Relief | 7 | 6 | 9
  4 Hours After Time 0: A Little Relief | 4 | 3 | 4
  4 Hours After Time 0: Some Relief | 0 | 2 | 1
  4 Hours After Time 0: A Lot of Relief | 3 | 4 | 1
  4 Hours After Time 0: Complete Relief | 1 | 0 | 0
  5 Hours After Time 0: No Relief | 8 | 8 | 9
  5 Hours After Time 0: A Little Relief | 2 | 3 | 5
  5 Hours After Time 0: Some Relief | 1 | 0 | 1
  5 Hours After Time 0: A Lot of Relief | 1 | 4 | 0
  5 Hours After Time 0: Complete Relief | 3 | 0 | 0
  6 Hours After Time 0: No Relief | 6 | 6 | 8
  6 Hours After Time 0: A Little Relief | 3 | 2 | 3
  6 Hours After Time 0: Some Relief | 0 | 3 | 3
  6 Hours After Time 0: A Lot of Relief | 4 | 3 | 1
  6 Hours After Time 0: Complete Relief | 2 | 1 | 0
  7 Hours After Time 0: No Relief | 6 | 5 | 8
  7 Hours After Time 0: A Little Relief | 2 | 1 | 2
  7 Hours After Time 0: Some Relief | 0 | 4 | 2
  7 Hours After Time 0: A Lot of Relief | 4 | 5 | 3
  7 Hours After Time 0: Complete Relief | 3 | 0 | 0
  8 Hours After Time 0: number analyzed (Participants) | 14 | 15 | 15
  8 Hours After Time 0: No Relief | 5 | 5 | 8
  8 Hours After Time 0: A Little Relief | 0 | 2 | 2
  8 Hours After Time 0: Some Relief | 3 | 4 | 1
  8 Hours After Time 0: A Lot of Relief | 4 | 3 | 4
  8 Hours After Time 0: Complete Relief | 2 | 1 | 0
  12 Hours After Time 0: number analyzed (Participants) | 13 | 15 | 15
  12 Hours After Time 0: No Relief | 3 | 2 | 2
  12 Hours After Time 0: A Little Relief | 1 | 2 | 4
  12 Hours After Time 0: Some Relief | 2 | 7 | 5
  12 Hours After Time 0: A Lot of Relief | 6 | 4 | 4
  12 Hours After Time 0: Complete Relief | 1 | 0 | 0
  16 Hours After Time 0: number analyzed (Participants) | 13 | 15 | 15
  16 Hours After Time 0: No Relief | 1 | 1 | 4
  16 Hours After Time 0: A Little Relief | 3 | 4 | 4
  16 Hours After Time 0: Some Relief | 2 | 3 | 6
  16 Hours After Time 0: A Lot of Relief | 5 | 6 | 1
  16 Hours After Time 0: Complete Relief | 2 | 1 | 0
  20 Hours After Time 0: number analyzed (Participants) | 13 | 15 | 15
  20 Hours After Time 0: No Relief | 1 | 1 | 1
  20 Hours After Time 0: A Little Relief | 4 | 2 | 2
  20 Hours After Time 0: Some Relief | 1 | 4 | 4
  20 Hours After Time 0: A Lot of Relief | 3 | 6 | 6
  20 Hours After Time 0: Complete Relief | 4 | 2 | 2
  24 Hours After Time 0: number analyzed (Participants) | 13 | 15 | 15
  24 Hours After Time 0: No Relief | 0 | 0 | 1
  24 Hours After Time 0: A Little Relief | 3 | 2 | 2
  24 Hours After Time 0: Some Relief | 2 | 3 | 4
  24 Hours After Time 0: A Lot of Relief | 6 | 9 | 6
  24 Hours After Time 0: Complete Relief | 2 | 1 | 2
  32 Hours After Time 0: number analyzed (Participants) | 13 | 14 | 15
  32 Hours After Time 0: No Relief | 1 | 0 | 2
  32 Hours After Time 0: A Little Relief | 3 | 2 | 3
  32 Hours After Time 0: Some Relief | 2 | 3 | 0
  32 Hours After Time 0: A Lot of Relief | 3 | 8 | 8
  32 Hours After Time 0: Complete Relief | 4 | 1 | 2
  40 Hours After Time 0: number analyzed (Participants) | 13 | 14 | 15
  40 Hours After Time 0: No Relief | 2 | 0 | 1
  40 Hours After Time 0: A Little Relief | 1 | 3 | 2
  40 Hours After Time 0: Some Relief | 2 | 5 | 4
  40 Hours After Time 0: A Lot of Relief | 3 | 5 | 7
  40 Hours After Time 0: Complete Relief | 5 | 1 | 1
  48 Hours After Time 0: number analyzed (Participants) | 13 | 14 | 15
  48 Hours After Time 0: No Relief | 1 | 0 | 1
  48 Hours After Time 0: A Little Relief | 2 | 4 | 0
  48 Hours After Time 0: Some Relief | 1 | 3 | 4
  48 Hours After Time 0: A Lot of Relief | 4 | 6 | 6
  48 Hours After Time 0: Complete Relief | 5 | 1 | 4

8. Secondary Outcome: Peak Pain Relief From Time 0 (First Dose of Study Medication)
Description: The highest level of pain relief achieved on a 5-point categorical scale where 0=none, 1=a little, 2=some, 3=a lot, 4=complete.
Time Frame: Within 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
Participants
  A Little Relief | 2 | 0 | 0
  Some Relief | 0 | 1 | 2
  A Lot of Relief | 5 | 11 | 7
  Complete Relief | 8 | 3 | 6

9. Secondary Outcome: Time (Minutes) to Peak Pain Relief From Time 0 (First Dose of Study Medication)
Time Frame: Within 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
minutes | 300.0 [30 to 955] | 420.0 [90 to 1198] | 1198 [45 to 1912]

10. Secondary Outcome: Time (Minutes) to First Perceptible Pain Relief From Time 0 (First Dose of Study Medication)
Description: Time to perceptible and meaningful pain relief will be evaluated using the 2-stopwatch method (after the first dose only) (2 stopwatches will be started as soon as the first dose of study drug is administered. Each participant will be instructed to stop the first stopwatch when he or she experiences any perceptible pain relief and the second stopwatch when he or she experiences pain relief that is meaningful to them.)
Time Frame: Within 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
minutes | 5 [2 to 15] | 10 [1 to 15] | 20 [3 to NA] — Not estimable because less than 50% of participants achieved perceptible pain relief.

11. Secondary Outcome: Time (Minutes) to Meaningful Pain Relief From Time 0 (First Dose of Study Medication)
Description: as for outcome 10
Time Frame: Within 48 hours after Time 0
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
minutes | 49 [10 to 87] | 190 [21 to NA] — Not estimable because less than 50% of participants achieved meaningful pain relief. | 79 [14 to NA] — Not estimable because less than 50% of participants achieved meaningful pain relief.

12. Secondary Outcome: Number of Participants Using Rescue Medication
Time Frame: Within 48 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Rescue Medication Used | 11 | 12 | 15
  No Rescue Medication Used | 4 | 3 | 0

13. Secondary Outcome: Time (Minutes) to First Use of Rescue Medication (Duration of Analgesia) Following Each Dose of the Investigational Product (IP)
Time Frame: Within 48 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
minutes | 204.0 [85 to 370] | 289.0 [98 to 431] | 126.0 [50 to 225]

14. Secondary Outcome: Number of Participants Using Rescue Analgesia Over 0 to 24 Hours and Over 0 to 48 Hours
Time Frame: Over 0 to 24 hours; Over 0 to 48 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Over 24 Hours | 11 | 12 | 15
  Over 48 hours | 11 | 12 | 15

15. Secondary Outcome: Participant Global Evaluation of Study Drug
Description: Participants provide a global evaluation of study drug on a 5-point categorical scale where 0=poor, 1=fair, 2=good, 3=very good, and 4=excellent.
Time Frame: Within 48 hours
Population: All randomized participants from the Intent-to-Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 15 | 15 | 15
Participants
  Poor | 2 | 3 | 4
  Fair | 3 | 2 | 0
  Good | 1 | 3 | 1
  Very Good | 3 | 3 | 8
  Excellent | 6 | 4 | 2

ADVERSE EVENTS:
Time Frame: Baseline up to 37 days approximately.
Arm/Group | Higher Dose Fentanyl Sublingual Spray | Lower Dose Fentanyl Sublingual Spray | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 12/15 | 8/15 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Dose Fentanyl Sublingual Spray (N=15) | Lower Dose Fentanyl Sublingual Spray (N=15) | Placebo (N=15)
Nausea (Gastrointestinal disorders) | 10 | 4 | 1
Vomiting (Gastrointestinal disorders) | 8 | 2 | 0
Application Site Pain (General disorders) | 3 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Burning Sensation (General disorders) | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal Mycotic Infection (Infections and infestations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Restless Leg Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 2 | 1
Headache (Nervous system disorders) | 4 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Oropharyngeal Swelling (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hot Flush (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-12-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT02915978/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT02915978/SAP_001.pdf